CLINICAL TRIAL: NCT06117410
Title: Assessing Ultrasonographic Severity of Adenomyosis - a Feasibility and Interobserver Study
Brief Title: Assessing Ultrasonographic Severity of Adenomyosis
Acronym: AdenoStaging
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, J.A.F. Huirne, Prof. Dr., Amsterdam UMC, location VUmc
Other Study IDs: 2021.0035
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Adenomyosis; Ultrasound
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this pilot study is to develop a feasible and quantifiable ultrasonographic method to grade the severity of adenomyosis and to determine the interobserver variation.

DETAILED DESCRIPTION:
The investigators will conduct a prospective observational study in premenopausal women visiting the gynaecological outpatient clinic for an ultrasonographic exam. Patients are recruited when the diagnosis adenomyosis was made with transvaginal ultrasound (TVUS). Diagnosis adenomyosis requires at least one direct US feature of adenomyosis (subendometrial lines or buds, hyperechogenic islands or myometrial cysts). The sonographers obtain two-dimensional (2D) images, a grey-scale video-clip, elastography and power-doppler and micro-vascularity flow clips and images, and a three-dimensional (3D) uterine volume. The investigators will evaluate the collected images, clips and 3D-volumes with different methods to assess severity and test the feasibility and inter-observer agreement of these methods.

At the outpatient clinic, all real-time TVUS are assessed in a systematically manner by the sonographers and the presence of MUSA (Morphological Uterus Sonographic Assessment) features (subendometrial lines or buds, hyperechogenic islands or myometrial cysts, asymmetrical myometrium, globular uterus, translesional vascularity, fan-shaped shadowing, interrupted/irregular junctional zone) and an estimation of the affected myometrium, graded in mild (<25% affected myometrium), moderate (25%-50% affected myometrium) or severe (>50% affected myometrium) are reported. Clinical data, medical history, reason for visit, pain score in numeric rating scale (NRS), pictorial blood assessment chart (PBAC) score, etc. is collected.

Based on previous research and experience, four experts in gynaecological sonography select multiple offline methods using 5D Viewer software, for the evaluation and quantification of the severity of adenomyosis.

All the ultrasounds will be coded, so the assessors are blinded for patients demographics, medical history, symptomatology and the assessment by the sonographers.

Two experienced gynaecologist and one resident in gynaecology will test these methods for feasibility. Feasibility will be scored regarding technique, time and interpretation of MUSA features. The selected feasible methods will be tested for inter-observer variation. Finally a comparison of the severity evaluation by the assessors done with the new methods and the results of the severity estimation at the outpatient clinic will be made.

The method(s) that obtained a good feasibility score and good inter-observer agreement will consecutively be used in a follow-up study investigating the correlation with symptomatology, e.g. pain (NRS) and PBAC score.

Additionally, a descriptive study using the elastography and micro-vascularity flow images and clips will be performed.

The obtained data will be analysed to determine a total feasibility score, inter-observer variation and inter-test agreement. Inter-observer variation was tested with Fleiss Kappa or Intra Class Correlation Coefficient (ICC), depending on the data used. A kappa-coefficient of 0.41-0.60 or an ICC value of 05.-0.75 was set as moderate, κ0.51-0.80 or ICC 0.75-0.9 as good and κ≥0.80 or ICC ≥0.9 as excellent agreement. A Jonckheere-Terpstra test was used to test the trend of the new severity score and the estimated assessment of MUSA. Inter-test agreement was calculated with Cohens weighted Kappa (κw). For the correlation with NRS and PBAC intraclass correlation and Fleiss kappa were calculated and the mean severity outcomes were correlated with NRS and PBAC.

All women will sign an informed consent.

ELIGIBILITY:
Inclusion Criteria:

* at least one direct MUSA feature (lines and buds, hyperechogenic islands, cysts)
* premenopausal, older than18 years

Exclusion Criteria:

* hormonal medication
* other reason for gynaecological symptoms, more evident than adenomyosis, e.g. deep infiltrating endometriosis, dominant uterine fibroids (>5cm, >5 myoma, intracavitary myoma), cervical or endometrial cancer.

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: Gynaecological premenopausal women visiting the outpatient clinic because of gynecololgical symptoms, older than 18 years, with sonographic signs of adenomyosis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Quantifiable offline severity method | Baseline
  Method using 5D viewer to assess severity of adenomyosis offline

SECONDARY OUTCOMES:
Dysmenorrhea | Baseline
  Painscore during menstruation, in numeric rating scale from respectively no pain to extreme pain (0-10)
Amount of menstrual blood loss | Baseline
  Evaluation of blood loss in pictorial blood assessment chart (PBAC). 0-150= normal bloodloss. >150= heavy menstrual bleeding.
Real-time severity estimation | Baseline
  Estimation of severity at outpatient clinic using MUSA features: mild (<25% affected myometrium), moderate (25-50% affected myometrium) or severe (>50% affected)
Numbers of MUSA features | Baseline
  Real-time presence of a number of individual MUSA features, as a measurement of severity of adenomyosis

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Van den Bosch T, de Bruijn AM, de Leeuw RA, Dueholm M, Exacoustos C, Valentin L, Bourne T, Timmerman D, Huirne JAF. Sonographic classification and reporting system for diagnosing adenomyosis. Ultrasound Obstet Gynecol. 2019 May;53(5):576-582. doi: 10.1002/uog.19096. No abstract available. PMID 29790217
- [Background] Harmsen MJ, Van den Bosch T, de Leeuw RA, Dueholm M, Exacoustos C, Valentin L, Hehenkamp WJK, Groenman F, De Bruyn C, Rasmussen C, Lazzeri L, Jokubkiene L, Jurkovic D, Naftalin J, Tellum T, Bourne T, Timmerman D, Huirne JAF. Consensus on revised definitions of Morphological Uterus Sonographic Assessment (MUSA) features of adenomyosis: results of modified Delphi procedure. Ultrasound Obstet Gynecol. 2022 Jul;60(1):118-131. doi: 10.1002/uog.24786. PMID 34587658